CLINICAL TRIAL: NCT02877303
Title: Phase II Study of the Hyper-CVAD Regimen in Sequential Combination With Blinatumomab With or Without Inotuzumab Ozogamicin as Frontline Therapy for Adults With B-Cell Lineage Acute Lymphocytic Leukemia
Brief Title: Blinatumomab, Inotuzumab Ozogamicin, and Combination Chemotherapy as Frontline Therapy in Treating Patients With B Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0845; NCI-2017-00596 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0845 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: B Acute Lymphoblastic Leukemia; B Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Inotuzumab Ozogamicin; Mercaptopurine; azathiopurine; Methotrexate; merphos; ofatumumab; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (blinatumomab, inotuzumab, combination chemotherapy) (Experimental): See detailed description.
  Interventions: Biological: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Biological: Inotuzumab Ozogamicin; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Biological: Ofatumumab; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Biological: Blinatumomab — Given IV
  Other Names: Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI-538; MT-103
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT and IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC-544; Way 207294; WAY-207294
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT, IV, and PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well blinatumomab, inotuzumab ozogamicin, and combination chemotherapy work as frontline therapy in treating patients with B acute lymphoblastic leukemia. Immunotherapy with monoclonal antibodies, such as blinatumomab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a toxic agent called ozogamicin. Inotuzumab attaches to CD22 positive cancer cells in a targeted way and delivers ozogamicin to kill them. Drugs used in chemotherapy, such as cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, dexamethasone, cytarabine, mercaptopurine, methotrexate, and prednisone work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving blinatumomab, inotuzumab ozogamicin, and combination chemotherapy may work better in treating patients with B acute lymphoblastic leukemia than chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the clinical efficacy of the sequential combination of hyperfractionated cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone (hyper-CVAD) + blinatumomab + inotuzumab ozogamicin (inotuzumab) in patients with newly diagnosed B-cell acute lymphoblastic leukemia (ALL) in terms of relapse-free survival (RFS).

SECONDARY OBJECTIVE:

I. To evaluate other efficacy endpoints such as overall survival, overall response rate, minimal residual disease (MRD) negativity rate as well as the safety of this combination.

EXPLORATORY OBJECTIVES:

I. To identify genomic alterations in adult ALL predictive for response and long-term outcomes with the combination of hyper-CVAD plus blinatumomab and inotuzumab.

II. To evaluate the impact of next generation sequencing (NGS)-based MRD assay on outcomes and to compare with standard flow cytometry MRD assays.

OUTLINE:

INTENSIVE PHASE: Patients receive cyclophosphamide intravenously (IV) over 3 hours twice daily (BID) on days 1-3, dexamethasone orally (PO) once daily (QD) on days 1-4 and 11-14, methotrexate intrathecally (IT) on day 2 of cycles 1 and 3, day 8 of cycles 2 and 4, and IV over 24 hours on day 1 of cycles 2 and 4, doxorubicin hydrochloride IV continuously on day 4, vincristine sulfate IV over 15 minutes on days 4 and 11, and cytarabine IT on day 7 of cycles 1 and 3, day 5 of cycles 2 and 4, and IV over 2 hours on days 2 and 3 of cycles 2 and 4. Patients may also receive ofatumumab IV or rituximab IV over 4-6 hours on days 1 and 11 of cycles 1 and 3, and days 1 and 8 of cycles 2 and 4 at the discretion of the treating physician. Patients may receive ofatumumab IV over 4-6 hours on day 2 of cycle 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

BLINATUMOMAB AND INOTUZUMAB OZOGAMICIN PHASE (CYCLES 5-8): Patients receive blinatumomab IV continuously on weeks 1-4. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 5 and 11 of cycles 6 and 8. Treatment repeats every 6 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: At doctor's discretion, patients may receive maintenance therapy prior to completing 4 cycles of hyper-CVAD and/or 4 cycles of blinatumomab. Patients receive mercaptopurine PO thrice daily (TID), methotrexate PO every week, vincristine sulfate IV over 15 minutes every month, and prednisone PO on days 1-5. Cycles repeat every 6 weeks for 12 months in the absence of disease progression or unacceptable toxicity. Patients also receive blinatumomab IV after every 3 cycles of maintenance therapy for a total of about 15 cycles.

After completion of study treatment, patients are followed up 1 time each month for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, previously untreated B-lineage ALL or lymphoblastic lymphoma, or having achieved complete remission (CR) with one course of induction chemotherapy; patients who require steroids, cytarabine (ara-c) or hydrea to manage disease symptoms prior to finalization of diagnosis and treatment plan are allowed and eligible
* Failure to one induction course of chemotherapy (these patients will be analyzed separately); patients who require steroids, ara-c or hydrea to manage disease symptoms prior to finalization of diagnosis and treatment plan are allowed and eligible
* Performance status of 0-3
* Creatinine less than or equal to 2.0 mg/dL (unless considered tumor related)
* Bilirubin less than or equal to 2.0 mg/dL (unless considered tumor related)
* Adequate cardiac function as assessed by history and physical examination
* No active or co-existing malignancy with life expectancy less than 12 months, sources for the determination of clinical significance by the treating physician will be included in the subject's medical record

Exclusion Criteria:

* Pregnant or nursing women
* Known to be human immunodeficiency virus (HIV)-positive
* Philadelphia chromosome (Ph)-positive ALL
* Active and uncontrolled disease/infection as judged by the treating physician, sources for the determination of clinical significance by the treating physician will be included in the subject's medical record
* Unable or unwilling to sign the consent form
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per treating physician assessment), sources for the determination of clinical significance by the treating physician will be included in the subject's medical record
* History or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis; (Patients with CNS involvement of leukemia are NOT excluded)
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement; auto-immune disease with possible CNS consequences/manifestations such as such as epilepsy, paresis, aphasia, stroke, dementia, Parkinson's disease, cerebellar disease, or psychosis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | From date of treatment start until the date of death or disease relapse, assessed for up to 24 months
  Will be estimated using the method of Kaplan and Meier. Will compute the Bayesian posterior probability. Will perform a competing risk analysis treating stem cell transplant as a competing event for RFS.

SECONDARY OUTCOMES:
Overall survival | Up to 24 months
  Will be estimated using the method of Kaplan and Meier.
Overall response rate | Up to 24 months
  Will be estimated along with the exact 95% confidence intervals.
Minimal residual disease negativity rate | Up to 24 months
  Will be estimated along with the exact 95% confidence intervals.
Incidence of adverse events | Up to 24 months
  Will be summarized by organ type, grade and attribution to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jabbour E, Short NJ, Jain N, Thompson PA, Kadia TM, Ferrajoli A, Huang X, Yilmaz M, Alvarado Y, Patel KP, Garcia-Manero G, Macaron W, Garris R, Konopleva M, Ravandi F, Kantarjian H. Hyper-CVAD and sequential blinatumomab for newly diagnosed Philadelphia chromosome-negative B-cell acute lymphocytic leukaemia: a single-arm, single-centre, phase 2 trial. Lancet Haematol. 2022 Dec;9(12):e878-e885. doi: 10.1016/S2352-3026(22)00285-X. Epub 2022 Oct 22. PMID 36279879
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- [Derived] Jabbour E, Kantarjian H. The Hyper-CVAD Regimen is an Optimal Pediatric-inspired Regimen for Adolescents and Adults With Acute Lymphoblastic Leukemia. Clin Lymphoma Myeloma Leuk. 2021 Jan;21(1):63-65. doi: 10.1016/j.clml.2020.09.001. Epub 2020 Oct 24. No abstract available. PMID 33191168
- See also: MD Anderson Cancer Center — http://www.mdanderson.org